CLINICAL TRIAL: NCT03210064
Title: A Phase II Clinical Trial Study on Apatinib and 5-Fu Combination Regimen in the Treatment of Advanced Colorectal Cancer Patients
Brief Title: Clinical Study of Apatinib and 5-Fu Combination Regimen to Treat Advanced Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui ting Xu，MD (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Hui ting Xu，MD, Deputy Chief Physician, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HXu
Record Dates: First submitted 2017-05-15; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Apatinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Experimental: apatinib combined with 5-Fu
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib and 5-Fluorouracil (Experimental): Apatinib 500 mg qd po.5-Fluorouracil 400mg/m2 iv d1，2400mg-3000mg/m2 civ 46h,q2w.5-Fluorouracil derivatives(Capecitabine 1000mg/m2 bid po d1-d14 q3w.S1 40mg/m2 bid po d1-d14 q3w).
  Interventions: Drug: Apatinib; Drug: 5-fluorouracil
- 5-Fluorouracil (Active Comparator): 5-Fluorouracil 400mg/m2 iv d1，2400mg-3000mg/m2 civ 46h,q2w.5-Fluorouracil derivatives(Capecitabine 1000mg/m2 bid po d1-d14 q3w.S1 40mg/m2 bid po d1-d14 q3w).
  Interventions: Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Apatinib — Apatinib Mesylate Tablets 500 mg qd po
  Other Names: 5-fluorouracil
  Arms: Apatinib and 5-Fluorouracil
Drug: 5-fluorouracil — 5-Fluorouracil 400mg/m2 iv d1，2400mg-3000mg/m2 civ 46h,q2w.5-Fluorouracil derivatives(Capecitabine 1000mg/m2 bid po d1-d14 q3w.S1 40mg/m2 bid po d1-d14 q3w).
  Other Names: 5-Fluorouracil derivatives

SUMMARY:
This study makes an observation over the objective response rate of Apatinib and 5-Fu combination regimen in the three-line treatment of metastatic colorectal cancer. All the participants will randomly receive the treatment of Apatinib and 5-Fu combination regimen or 5-Fu.

DETAILED DESCRIPTION:
5-Fu chemotherapy is an effective therapy for colorectal cancer. Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular endothelial growth factor receptor 2 (VEGFR-2), with a decrease in VEGF-mediated endothelial cell migration, proliferation, and tumor microvascular density. A phase II trail of Apatinib has been demonstrated that Apatinib is safe to treat the metastatic colorectal cancer and the disease control rate can reach 50%.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤ 70 years of age

  * Histological confirmed advanced or metastatic colorectal Cancer，at least one measurable lesion, larger than 10 mm in diameter by spiral CT scan(scanning layer ≤ 5 mm )
  * Have failed for ≥ 2 lines of chemotherapy
  * Life expectancy of more than 3 months
  * ECOG performance scale ≤ 1
  * Duration from the last therapy is more than 6 weeks for nitroso or mitomycin More than 4 weeks for operation, radiotherapy or cytotoxic agents
  * Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 × 10E+9/L, neutrophil > 1.5 × 10E+9/L, serum creatinine ≤ 1×upper limit of normal(ULN), bilirubin < 1.25 ULN, and serum transaminase ≤ 2.5× ULN)
  * Child bearing potential, a negative urine or serum pregnancy test result before initiating apatinib, must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article.
  * Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite using single medical therapy, more than class I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia(including QTcF:male ≥ 450 ms, female ≥ 470 ms), or cardiac insufficiency myocardial ischemia, arrhythmia, or cardiac insufficiency
* Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Any factors that influence the usage of oral administration Evidence of CNS metastasis
* URT: urine protein ≥ (++)and > 1.0 g of 24 h
* PT, APTT, TT, Fbg abnormal, having hemorrhagic tendency (eg. active peptic ulcer disease) or receiving the therapy of thrombolysis or anticoagulation
* Abuse of drugs
* Certain possibility of gastric or intestine hemorrhage
* Less than 4 weeks from the last clinical trial
* Viral hepatitis type B or type C
* Prior VEGFR inhibitor treatment
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-04-24 (Estimated); Study Completion 2019-04-24 (Estimated)

PRIMARY OUTCOMES:
ORR | From assignment of the first subject to 3 months later after the last participant is recruited.
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)

SECONDARY OUTCOMES:
DCR | From assignment of the first subject to 3 months later after the last participant is recruited.
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)
PFS | From assignment of the first subject to 3 months later after the last participant is recruited.
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
OS | From assignment of the first subject until 30 death events observed, up to 2 years.
  OS is defined as the time from date of assignment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
QoL | From assignment of the first subject to 3 months later after the last participant is recruited.
  The general well-being of participants, outlining negative and positive features of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yan li Nie, MD, Principal Investigator — Hu bei CH; Liu Yang, MD, Study Director — Hu bei CH
Locations (1):
- Hui ting Xu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen R, Yang L, Hu S, Yin Z, Nie Y, Xu H, Zhong Y, Zhu Y, Liang X, Xu H. Apatinib plus 5-fluorouracil as a third or subsequent-line treatment option for metastatic colorectal cancer: a phase-II, single-arm, prospective study. Ann Transl Med. 2022 Jan;10(2):100. doi: 10.21037/atm-22-77. PMID 35282086